CLINICAL TRIAL: NCT04507321
Title: A Two-period Study in Healthy Male Participants to Determine the Pharmacokinetics, Balance/Excretion, and Metabolism of [14C]-GSK3640254 Following a Single Intravenous Radiolabeled Microtracer Dose (Concomitant With a Non-radiolabeled Oral Dose) and a Single Oral Radiolabeled Dose
Brief Title: Pharmacokinetics and Metabolism of 14 Carbon [14C]-GSK3640254
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213051; 2019-004444-30 (EudraCT Number)
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Results first posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-11

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus (HIV); GSK3640254; Pharmacokinetics; Radiolabeled; Mass balance
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — GSK3640254

STUDY DESIGN:
Intervention Model Description: Participants will receive non-radiolabeled GSK3640254 oral tablets concomitantly with radiolabeled [14C]-GSK3640254 administered as an IV infusion in treatment Period 1 and radiolabeled [14C]-GSK3640254 as an oral suspension in treatment Period 2.
Masking Description: This will be an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GSK3640254 tablet + [14C]-GSK3640254 IV/[14C] oral suspension (Experimental): Participants will receive a single oral dose of GSK3640254 200 milligram (mg) (2×100 mg) tablets with a moderate fat meal. Participants will then be administered a 100 microgram (mcg) dose (approximately 3.7 kilobecquerel; 100 nano Curie) of [14C]-GSK3640254 as an IV infusion for 1 hour on Day 1 in treatment Period 1, On Day 1 in treatment Period 2, participants will receive a single oral dose of 85 mg (approximately 3.15 megabecquerel; 85 micro Curie) [14C]-GSK3640254 administered as an oral suspension with a moderate fat meal. A wash out period of at least 13 days will be maintained between oral doses of treatment periods.
  Interventions: Drug: GSK3640254 Oral tablet; Drug: [14C]-GSK3640254 intravenous infusion; Drug: [14C]-GSK3640254 powder

INTERVENTIONS:
Drug: GSK3640254 Oral tablet — GSK3640254 will be available as white film-coated round tablets to be administered via oral route with meal in the morning with 240 milliliter (mL) of water at room temperature.
Drug: [14C]-GSK3640254 intravenous infusion — [14C]-GSK3640254 will be available as clear, colorless solution free from visible particulates to be administered via the IV route.
Drug: [14C]-GSK3640254 powder — [14C]-GSK3640254 will be available as white powder to be reconstituted into a suspension with 25 mL of vehicle before dosing so as to administer 85 mg dose with meal in the morning.

SUMMARY:
This is an open-label, single-center, single group, non-randomized, two-period, single sequence, mass balance study which will enroll 6 healthy male participants. This study will assess the pharmacokinetics, balance/excretion, and metabolism of GSK3640254 in humans using [14C]-radiolabeled drug substance administered as an intravenous (IV) infusion and via the oral route. The study will also provide an assessment of GSK3640254 absorption, metabolism and excretion following administration of a [14C]-radiolabeled oral suspension. Each participant will be involved in the study for up to 10 weeks which will include a screening period, two treatment periods (treatment Periods 1 and 2) separated by a washout of at least 13 days between oral doses, and a follow-up visit 7-14 days after the last assessment in treatment Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 30 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and ECG. A participant with a clinical abnormality or laboratory parameter (i.e. outside the reference range for the population being studied), which is not specifically listed in the eligibility criteria, may be included only if the investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* History of regular bowel movements (averaging one or more bowel movements per day).
* Non-smoker, or ex-smoker who hasn't regularly smoked for the 6 months before Screening.
* Body weight of 50 kilograms (kg) and above, and body mass index (BMI) within the range 19.0 to 31.0 kg/square meter (m^2) (inclusive).
* Male participants are eligible to participate if they agree to the following during the study, including washout periods: Refrain from donating sperm and either a) be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or b) Agree to use a male condom when having penile-vaginal intercourse with a woman of childbearing potential unless vasectomized.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Participants with a history of cholecystectomy must be excluded.
* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Any clinically relevant abnormality identified at the Screening medical assessment (physical examination/medical history) clinical laboratory tests, or 12-lead ECG.
* Current episode, recent history, or chronic history of diarrhea.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Any history of significant underlying psychiatric disorder, including, but not limited to, schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment. Participants with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the ViiV Healthcare (VH)/GlaxoSmithKline (GSK) Medical Monitor.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the participant's ability to comply with the dosing schedule and protocol.
* Regular use of known drugs of abuse or history of drug abuse or dependence within 6 months of the study.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 grams of alcohol: a glass (equivalent to [~]240 mL) of beer, 1 small glass (~100 mL) of wine or 1 (~25 mL) measure of spirits.
* History of or regular use of tobacco- or nicotine-containing products in the 3 months prior to Screening.
* Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.
* QT duration corrected for heart rate by Fridericia's formula (QTcF) >450 milliseconds (msec).
* At Screening or prior to the first dose, a supine blood pressure (BP) that is persistently higher than 140/90 millimeters of mercury (mmHg).
* At Screening or prior to the first dose, a supine mean heart rate (HR) outside the range of 50 to 100 beats per minute (bpm). A heart rate from 100 to 110 bpm can be rechecked by ECG or vital signs within 30 minutes to verify eligibility.
* A participant with known or suspected active COVID-19 infection OR contact with an individual with known COVID-19, within 14 days of study enrollment.
* Past or intended use of over-the-counter or prescription medication, including analgesics (example [e.g], paracetamol), herbal medications, or grapefruit and Seville orange juices within 14 days prior to the first dose of study intervention until completion of the follow-up visit unless approved by the Investigator in conjunction with a VH/GSK Medical monitor.
* Treatment with any vaccine within 30 days prior to receiving study intervention.
* Current enrollment in a clinical trial; recent participation in a clinical trial and has received an investigational product within 3 months before the first dose in the current study.
* Exposure to more than 4 new chemical entities within 12 months before the first dose in the current study.
* Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months. A participant's previous effective dose will be reviewed by the medical investigator to ensure there is no risk of contamination/carryover into the current study.
* Received a total body radiation dose of greater than 10.0 millisievert (mSv) (upper limit of International Commission on Radiological Protection [ICRP] category II) or exposure to significant radiation (e.g., serial x-ray or computed tomography [CT] scans, barium meal, etc.) in the 3 years before this study.
* Alanine transaminase (ALT) >=1.5 times upper limit of normal (ULN). A single repeat of ALT is allowed within a single Screening period to determine eligibility.
* Bilirubin >=1.5 times ULN (isolated bilirubin >=1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent (%). A single repeat of any laboratory abnormality is allowed within a single Screening period to determine eligibility.
* Presence of Hepatitis B surface antigen (HBsAg) at Screening or positive Hepatitis C antibody test result at Screening or within 3 months before the first dose of study intervention and positive on reflex to hepatitis C ribonucleic acid (RNA).
* Positive HIV-1 and -2 antigen/antibody immunoassay at Screening.
* Any positive (abnormal) response confirmed by the investigator or qualified designee-administered Columbia-Suicide Severity Rating Scale (C-SSRS).
* Any Grade 2 to 4 laboratory abnormality at Screening, with the exception of creatine phosphokinase (CPK) and lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT (described above), will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any laboratory abnormality (other than a viral Screening test for HIV-1/2, hepatitis B Virus [HBV], or hepatitis C Virus [HCV]) is allowed within a single Screening period to determine eligibility.
* Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction in the past 3 months, symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, non-sustained or sustained ventricular tachycardia, second-degree atrioventricular block Mobitz Type II, third-degree atrioventricular block, complete heart block, or conduction abnormality) which, in the opinion of the investigator or VH/GSK Medical Monitor, will interfere with the safety for the individual participant. Any acute laboratory abnormality at Screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Has had an occupation which requires monitoring for radiation exposure, nuclear medicine procedures, or excessive x-rays within the past 3 years.
* Loss of more than 400 mL blood during the 3 months before Screening, e.g., as a blood donor, or plan to donate blood or blood products in the 3 months after the end of the trial.
* Unwillingness or inability to follow the procedures outlined in the protocol, including the use of the string bile collection device.
* History of sensitivity to GSK3640254, or their components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male participants will be part of this study.
Enrollment: 5 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, non-randomized, 2-period, single-sequence study to determine the pharmacokinetics, balance/excretion, and metabolism of radiolabeled [14C]-GSK3640254 following a single intravenous radiolabeled microtracer dose and a single oral radiolabeled dose. The study was conducted at a single center in the United Kingdom.
Pre-assignment Details: A total of 5 participants were enrolled in the study. The washout time between dosing in consecutive study periods was at least 13 days.
Groups:
- GSK3640254 Tablet+[14C]-GSK3640254 IV/ [14C]-GSK3640254 Oral Suspension: Participants were administered a single oral dose of GSK3640254 200 milligram (mg) (2×100 mg) tablets with a moderate fat meal, followed by an intravenous (IV) infusion of [14C]-GSK3640254 100 micrograms for 1 hour on Day 1 in Treatment Period 1. In Treatment Period 2 on Day 1, participants were administered a single oral dose of 85 mg [14C]-GSK3640254 as an oral suspension with a moderate fat meal. The treatment periods were separated by a washout period of at least 13 days between oral doses.
Period: Treatment Period 1 (8 Days)
Arm/Group | GSK3640254 Tablet+[14C]-GSK3640254 IV/ [14C]-GSK3640254 Oral Suspension
Started | 5
Completed | 5
Not Completed | 0
Period: Treatment Period 2 (8 Days)
Arm/Group | GSK3640254 Tablet+[14C]-GSK3640254 IV/ [14C]-GSK3640254 Oral Suspension
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GSK3640254 Tablet+[14C]-GSK3640254 IV/ [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.4 (5.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian- Central/South Asian Heritage | 1
  Black or African American | 3
  White- White/Caucasian/European Heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) in Plasma Following Administration of Oral Dose of GSK3640254
Description: Blood samples were collected at the indicated time points for Pharmacokinetic (PK) analysis. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.25, 5.5, 6, 7, 8, 9, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population comprised of all participants in the Safety Population (all participants who took atleast one dose of study intervention) who had at least 1 non-missing PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- GSK3640254 Tablet: Eligible participants received a single oral dose of 200 milligram (mg) (2×100 mg) tablets with a moderate fat meal on Day 1 in treatment Period 1
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Hours*nanogram per milliliter | 41234.1841 (14.5)

2. Primary Outcome: AUC(0-inf) of Total Radioactivity in Blood Following Administration of Oral Dose of GSK3640254
Description: Blood samples were collected at indicated time points. Data was not collected because a discrepancy has been identified in the Objectives and Endpoints section of the Protocol, which incorrectly states one of the Primary Endpoints. The Objectives and Endpoints section incorrectly states that the PK parameters of both the parent and total drug-related material (radioactivity) in plasma and blood would be presented. Neither the Schedule of Activities nor the Study Assessments and Procedures sections of the Protocol address the sampling and measurement of concentrations of parent drug in blood or calculation of derived PK parameters. Consequently, no parent analyte measurements were performed for blood samples. Thus, the reference to parent analyte specifically for blood, in the Objectives and Endpoints section was an error. Only samples and measurements for total drug-related material (radioactivity) in blood and plasma, and parent drug in plasma were collected to derive PK parameters.
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram Equivalent per milliliter
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Hours*nanogram Equivalent per milliliter | NA (NA) — Not applicable (NA) indicates data was not collected for this outcome measure as it was incorrectly stated as one of the Primary Endpoint in Objectives and Endpoints section of the Protocol, where the reference to parent analyte specifically for blood was an error. Only samples and measurements for total drug-related material (radioactivity) in blood and plasma, and parent drug in plasma were collected to derive PK parameters.

3. Primary Outcome: AUC(0-inf) in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- [14C]-GSK3640254 IV: Eligible participants received an intravenous (IV) infusion of [14C]-GSK3640254 100 micrograms for 1 hour on Day 1 in treatment Period 1.
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Hours*nanogram per milliliter | 96.5532 (19.7)

4. Primary Outcome: AUC(0-inf) of Total Radioactivity in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram Equivalent per milliliter
Groups:
- [14C]-GSK3640254 IV: Eligible participants received an IV infusion of [14C]-GSK3640254 100 micrograms for 1 hour on Day 1 in treatment Period 1
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Hours*nanogram Equivalent per milliliter | 105.0882 (19.1)

5. Primary Outcome: AUC(0-inf) in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- [14C]-GSK3640254 Oral Suspension: Eligible participants received a single oral dose of 85 mg [14C]-GSK3640254 as an oral suspension with a moderate fat meal on Day 1 in treatment period 2
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours*nanogram per milliliter | 19026.4818 (21.8)

6. Primary Outcome: AUC(0-inf) of Total Radioactivity in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram Equivalent per milliliter
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours*nanogram Equivalent per milliliter | 23226.8511 (20.7)

7. Primary Outcome: AUC(0-inf) of Total Radioactivity in Blood Following Administration of Oral Dose of [14C]-GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis. Data was not collected for this Outcome measure as AUC(0-inf) is not calculable for total radioactivity in blood due to insufficient sampling in the terminal phase.
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram Equivalent per milliliter
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours*nanogram Equivalent per milliliter | NA (NA) — NA indicates data was not collected for this outcome measure as AUC(0-inf) is not calculable for total radioactivity in blood due to insufficient sampling in the terminal phase.

8. Primary Outcome: AUC From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC[0-t]) in Plasma Following Administration of Oral Dose of GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- GSK3640254 Tablet: Eligible participants received a single oral dose of 200 mg (2×100 mg) tablets with a moderate fat meal on Day 1 in treatment Period 1
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Hours*nanogram per milliliter | 40816.9451 (14.2)

9. Primary Outcome: AUC(0-t) of Total Radioactivity in Blood Following Administration of Oral Dose of GSK3640254
Description: as for outcome 2
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram Equivalent per milliliter
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Hours*nanogram Equivalent per milliliter | NA (NA) — NA indicates data was not collected for this outcome measure as it was incorrectly stated as one of the Primary Endpoint in Objectives and Endpoints section of the Protocol, where the reference to parent analyte specifically for blood was an error. Only samples and measurements for total drug-related material (radioactivity) in blood and plasma, and parent drug in plasma were collected to derive PK parameters.

10. Primary Outcome: AUC(0-t) in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Hours*nanogram per milliliter | 93.3371 (20.4)

11. Primary Outcome: AUC(0-t) of Total Radioactivity in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram Equivalent per milliliter
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Hours*nanogram Equivalent per milliliter | 101.8025 (19.4)

12. Primary Outcome: AUC (0-t) in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours*nanogram per milliliter | 18828.0326 (21.7)

13. Primary Outcome: AUC(0-t) of Total Radioactivity in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram Equivalent per milliliter
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours*nanogram Equivalent per milliliter | 22746.1486 (20.4)

14. Primary Outcome: AUC(0-t) of Total Radioactivity in Blood Following Administration of Oral Dose of [14C]-GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram Equivalent per milliliter
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours*nanogram Equivalent per milliliter | 2395.2833 (17.7)

15. Primary Outcome: Maximum Observed Concentration (Cmax) in Plasma Following Administration of Oral Dose of GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Nanogram per milliliter | 1293.0 (7.6)

16. Primary Outcome: Cmax of Total Radioactivity in Blood Following Administration of Oral Dose of GSK3640254
Description: as for outcome 2
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram Equivalent per milliliter
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Nanogram Equivalent per milliliter | NA (NA) — NA indicates data was not collected for this outcome measure as it was incorrectly stated as one of the Primary Endpoint in Objectives and Endpoints section of the Protocol, where the reference to parent analyte specifically for blood was an error. Only samples and measurements for total drug-related material (radioactivity) in blood and plasma, and parent drug in plasma were collected to derive PK parameters.

17. Primary Outcome: Cmax in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Nanogram per milliliter | 8.435 (12.0)

18. Primary Outcome: Cmax of Total Radioactivity in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram Equivalent per milliliter
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Nanogram Equivalent per milliliter | 7.462 (6.9)

19. Primary Outcome: Cmax in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Nanogram per milliliter | 628.2 (15.4)

20. Primary Outcome: Cmax of Total Radioactivity in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram Equivalent per milliliter
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Nanogram Equivalent per milliliter | 675.312 (13.6)

21. Primary Outcome: Cmax of Total Radioactivity in Blood Following Administration of Oral Dose of [14C]-GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram Equivalent per milliliter
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Nanogram Equivalent per milliliter | 377.5 (23.9)

22. Primary Outcome: Time of Occurrence of Cmax (Tmax) in Plasma Following Administration of Oral Dose of GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Hours | 7.00 [4.5 to 9.0]

23. Primary Outcome: Tmax of Total Radioactivity in Blood Following Administration of Oral Dose of GSK3640254
Description: as for outcome 2
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Hours | NA [NA to NA] — NA indicates data was not collected for this outcome measure as it was incorrectly stated as one of the Primary Endpoint in Objectives and Endpoints section of the Protocol, where the reference to parent analyte specifically for blood was an error. Only samples and measurements for total drug-related material (radioactivity) in blood and plasma, and parent drug in plasma were collected to derive PK parameters.

24. Primary Outcome: Tmax in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Hours | 0.983 [0.983 to 0.983]

25. Primary Outcome: Tmax of Total Radioactivity in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Hours | 0.983 [0.983 to 0.983]

26. Primary Outcome: Tmax in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours | 4.00 [1.5 to 5.5]

27. Primary Outcome: Tmax of Total Radioactivity in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours | 4.0000 [1.500 to 6.000]

28. Primary Outcome: Tmax of Total Radioactivity in Blood Following Administration of Oral Dose of [14C]-GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours | 6.0 [2 to 10]

29. Primary Outcome: Terminal Phase Half-life (T1/2) in Plasma Following Administration of Oral Dose of GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Hours | 24.0860 (16.4)

30. Primary Outcome: T1/2 of Total Radioactivity in Blood Following Administration of Oral Dose of GSK3640254
Description: as for outcome 2
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Hours | NA (NA) — NA indicates data was not collected for this outcome measure as it was incorrectly stated as one of the Primary Endpoint in Objectives and Endpoints section of the Protocol, where the reference to parent analyte specifically for blood was an error. Only samples and measurements for total drug-related material (radioactivity) in blood and plasma, and parent drug in plasma were collected to derive PK parameters.

31. Primary Outcome: T1/2 in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Hours | 21.6959 (12.6)

32. Primary Outcome: T1/2 of Total Radioactivity in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Hours | 29.7527 (11.3)

33. Primary Outcome: T1/2 in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours | 24.2493 (5.1)

34. Primary Outcome: T1/2 of Total Radioactivity in Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours | 30.0505 (11.4)

35. Primary Outcome: T1/2 of Total Radioactivity in Blood Following Administration of Oral Dose of [14C]-GSK3640254
Description: Blood samples were collected at indicated time points for PK analysis. Data was not collected for this Outcome measure as T1/2 is not calculable for total radioactivity in blood due to insufficient sampling in the terminal phase.
Time Frame: Day 1: 2, 4, 6, 8, 10 hours
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Hours | NA (NA) — NA indicates data was not collected for this outcome measure as T1/2 is not calculable for total radioactivity in blood due to insufficient sampling in the terminal phase.

36. Primary Outcome: Volume of Distribution at Steady State (Vss) in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Liters | 28.7435 (21.9)

37. Primary Outcome: Clearance (CL) in Plasma Following Administration of IV Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Liters per hour | 1.0357 (19.7)

38. Primary Outcome: Renal Clearance (CLr) Following Administration of IV Dose of [14C]-GSK3640254
Description: Blood samples were collected at the indicated time points for PK analysis. Renal clearance was calculated as (Cumulative amount [Ae][Urine] for Period 1)/(Plasma AUC[0-inf]).
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Liters per hour | 0.01992 (29.2)

39. Primary Outcome: CLr Following Administration of Oral Dose of [14C]-GSK3640254
Description: Blood samples were collected at the indicated time points for PK analysis. Renal clearance was calculated as (Cumulative Ae[Urine] for Period 2)/(Plasma AUC[0-inf]).
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Liters per hour | 0.01465 (30.1)

40. Primary Outcome: Oral Clearance (CL/F) in Plasma Following Administration of Oral Dose of GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Liters per hour | 4.8503 (14.5)

41. Primary Outcome: CL/F in Plasma Following Administration Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Liters per hour | 4.4675 (21.8)

42. Primary Outcome: Apparent Volume of Distribution (Vz/F) Following Administration of Oral Dose of GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | GSK3640254 Tablet
Number analyzed (Participants) | 5
Liters | 168.5433 (14.0)

43. Primary Outcome: Vz/F Following Administration of Oral Dose of [14C]-GSK3640254
Description: as for outcome 3
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Liters | 156.2909 (19.0)

44. Primary Outcome: Absolute Oral Bioavailability of GSK3640254
Description: Absolute bioavailability is the amount of drug from a formulation that reaches the systemic circulation relative to an IV dose, computed as ratio of AUC(Oral Tablet)/Dose(Oral Tablet) with AUC(IV)/Dose(IV). Plasma samples were collected from participants at indicated time points. Absolute bioavailability from the oral tablet and IV doses were analyzed using AUC(0-inf) and AUC(0-t) pharmacokinetic parameters.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of dose normalized AUC
Groups:
- GSK3640254 Tablet + [14C]-GSK3640254 IV: Eligible participants were administered a single oral dose of GSK3640254 200 mg (2×100 mg) tablets with a moderate fat meal, followed by an IV infusion of [14C]-GSK3640254 100 micrograms for 1 hour on Day 1 in Treatment Period 1.
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Ratio of dose normalized AUC
  AUC (0 to infinity) | 0.2317 (10.1)
  AUC (0 to t) | 0.2373 (11.1)

45. Primary Outcome: Percentage of Drug Escaping First Pass Hepatic Clearance (Fh) Following Administration of [14C]-GSK3640254 IV
Description: Blood samples were collected at the indicated time points for PK analysis. Fh was expressed as percentage and was calculated as: 1 minus hepatic extraction ratio multiplied by 100. Hepatic extraction ratio=hepatic blood clearance (milliliters per minute)/hepatic blood flow (milliliters per minute).
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of drug escaped
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Percentage of drug escaped | 0.9945 (0.1)

46. Primary Outcome: Percentage of Drug Absorbed (Fa) Following Administration of [14C]-GSK3640254 Oral Suspension
Description: Blood samples were collected at the indicated time points for PK analysis. Fa was expressed as percentage which was calculated as ratio of oral bioavailability and Fh multiplied by 100.
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of drug absorbed
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Percentage of drug absorbed | 0.2595 (8.9)

47. Primary Outcome: Percentage of Drug Escaping Gut Metabolism (Fg) Following Administration of [14C]-GSK3640254 Oral Suspension
Description: Blood samples were collected at the indicated time points for PK analysis. Fg is defined as the fraction metabolized by gut wall as a fraction of the oral dose and was expressed as 1 minus Metabolite load following intravenous and oral administration multiplied by 100.
Time Frame: Day 1 (Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of drug escaped
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Percentage of drug escaped | 0.8980 (5.5)

48. Primary Outcome: Percentage of Total Radioactive Dose Excreted in Urine Following Administration of IV Dose of [14C]-GSK3640254
Description: Urine samples were collected at indicated timepoints to measure percentage of the total radioactive drug-related material excreted in urine. Percentage of radioactive dose excreted in urine was calculated as (amount excreted in urine divided by administered radioactivity dose) multiplied by 100. Not applicable (NA) indicates that No concentration values detected for pre-dose.
Time Frame: Day 1 (Pre-dose), 5, 24, 48, 72, 96, 120, 144 and 163 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Percentage of dose excreted
  Pre-dose | NA (NA) — No concentration values detected for pre-dose.
  5 hours | 0 (0.514)
  24 hours | 1.1 (0.382)
  48 hours | 1.61 (0.514)
  72 hours | 1.76 (0.551)
  96 hours | 1.82 (0.577)
  120 hours | 1.84 (0.581)
  144 hours | 1.85 (0.585)
  163 hours | 1.86 (0.589)

49. Primary Outcome: Percentage of Total Radioactive Dose Excreted in Urine Following Administration of Oral Dose of [14C]-GSK3640254
Description: Urine samples were collected at indicated timepoints to measure percentage of the total radioactive drug-related material excreted in urine. Percentage of radioactive dose excreted in urine was calculated as (amount excreted in urine divided by administered radioactivity dose) multiplied by 100.
Time Frame: Day 1 (Pre-dose), 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 and 288 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Percentage of dose excreted
  Pre-dose | 0.00 (0.00)
  24 hours | 0.14 (0.03)
  48 hours | 0.26 (0.06)
  72 hours | 0.31 (0.08)
  96 hours | 0.33 (0.11)
  120 hours | 0.34 (0.12)
  144 hours | 0.35 (0.13)
  168 hours | 0.35 (0.13)
  192 hours | 0.35 (0.13)
  216 hours | 0.35 (0.13)
  240 hours | 0.35 (0.13)
  264 hours | 0.35 (0.13)
  288 hours | 0.35 (0.13)

50. Primary Outcome: Percentage of Total Radioactive Dose Excreted in Feces Following Administration of IV Dose of [14C]-GSK3640254
Description: Fecal samples were collected at indicated timepoints to measure percentage of the total radioactive drug-related material excreted in feces. Percentage of radioactive dose excreted was calculated as (amount excreted in feces homogenate divided by administered radioactivity dose) multiplied by 100. NA indicates that No concentration values detected for pre-dose.
Time Frame: Day 1 (Pre-dose), 24, 48, 72, 96, 120, 144 and 163 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted
Arm/Group | [14C]-GSK3640254 IV
Number analyzed (Participants) | 5
Percentage of dose excreted
  Pre-dose | NA (NA) — No concentration values detected for pre-dose.
  24 hours | 0.0855 (0.0690)
  48 hours | 14.6 (9.40)
  72 hours | 41.7 (13.2)
  96 hours | 52.0 (12.1)
  120 hours | 61.1 (6.67)
  144 hours | 72.1 (5.76)
  163 hours | 73.6 (4.87)

51. Primary Outcome: Percentage of Total Radioactive Dose Excreted in Feces Following Administration of Oral Dose of [14C]-GSK3640254
Description: Fecal samples were collected at indicated timepoints to measure percentage of the total radioactive drug-related material excreted in feces. Percentage of radioactive dose excreted was calculated as (amount excreted in feces homogenate divided by administered radioactivity dose) multiplied by 100.
Time Frame: Day 1 (Pre-dose), 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 and 288 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Percentage of dose excreted
  Pre-dose | 0.00 (0.00)
  24 hours | 0.38 (0.59)
  48 hours | 37.8 (35.1)
  72 hours | 62.8 (35.9)
  96 hours | 71.0 (37.5)
  120 hours | 81.9 (38.3)
  144 hours | 86.8 (42.4)
  168 hours | 89.9 (42.6)
  192 hours | 90.0 (42.3)
  216 hours | 90.5 (43.0)
  240 hours | 90.5 (43.0)
  264 hours | 90.7 (43.3)
  288 hours | 90.8 (43.4)

52. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with common (greater than or equal to [>=]5 percent [%]) non-serious AEs and SAEs is presented.
Time Frame: Up to 50 days
Population: Safety Population comprised of all participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Participants
  Any Non-serious AEs | 1 | 1
  Any SAEs | 0 | 0

53. Secondary Outcome: Number of Participants With Worst Case Hematology Results Relative to Normal Range Post Baseline Relative to Baseline
Description: Blood samples were collected to analyze following hematology parameters; Basophils, Eosinophils, Erythrocytes mean corpuscular hemoglobin (MCH), Erythrocytes mean corpuscular volume (MCV), Erythrocytes, Hematocrit (HCT), Hemoglobin (Hb), Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets, Reticulocytes and Reticulocytes/Erythrocytes. Participants were counted in worst case category if their value changed to (low, normal or high), unless there was no change in their category. Participants whose laboratory value category was unchanged (for example [e.g.] High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Baseline value=latest pre-dose assessment (prior to the oral dose) in each treatment period, with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1: pre-dose) and Up to 50 Days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Participants
  Basophils, To Low | 0 | 0
  Basophils, To Normal or No Change | 5 | 5
  Basophils, To High | 0 | 0
  Eosinophils, To Low | 0 | 0
  Eosinophils, To Normal or No Change | 5 | 5
  Eosinophils, To High | 0 | 0
  Erythrocytes MCH, To Low | 0 | 0
  Erythrocytes MCH, To Normal or No Change | 5 | 5
  Erythrocytes MCH, To High | 0 | 0
  Erythrocytes MCV, To Low | 0 | 0
  Erythrocytes MCV, To Normal or No Change | 5 | 5
  Erythrocytes MCV, To High | 0 | 0
  Erythrocytes, To Low | 0 | 0
  Erythrocytes, To Normal or No Change | 5 | 5
  Erythrocytes, To High | 0 | 0
  Hematocrit, To Low | 0 | 2
  Hematocrit, To Normal or No Change | 5 | 3
  Hematocrit, To High | 0 | 0
  Hemoglobin, To Low | 0 | 1
  Hemoglobin, To Normal or No Change | 5 | 4
  Hemoglobin, To High | 0 | 0
  Leukocytes, To Low | 0 | 0
  Leukocytes, To Normal or No Change | 5 | 5
  Leukocytes, To High | 0 | 0
  Lymphocytes, To Low | 0 | 0
  Lymphocytes, To Normal or No Change | 5 | 5
  Lymphocytes, To High | 0 | 0
  Monocytes, To Low | 0 | 0
  Monocytes, To Normal or No Change | 5 | 5
  Monocytes, To High | 0 | 0
  Neutrophils, To Low | 0 | 0
  Neutrophils, To Normal or No Change | 5 | 5
  Neutrophils, To High | 0 | 0
  Platelets, To Low | 0 | 0
  Platelets, To Normal or No Change | 5 | 4
  Platelets, To High | 0 | 1
  Reticulocytes, To Low | 0 | 0
  Reticulocytes, To Normal or No Change | 4 | 5
  Reticulocytes, To High | 1 | 0
  Reticulocytes/Erythrocytes, To Low | 0 | 0
  Reticulocytes/Erythrocytes, To Normal or No Change | 4 | 5
  Reticulocytes/Erythrocytes, To High | 1 | 0

54. Secondary Outcome: Number of Participants With Worst Case Clinical Chemistry Results Relative to Normal Range Post Baseline Relative to Baseline
Description: Blood samples were collected to analyze following clinical chemistry parameters:Alanine aminotransferase(ALT),albumin,alkaline phosphatase(ALP),aspartate aminotransferase(AST),bilirubin,calcium,chloride,cholesterol,creatinine,direct bilirubin,globulin,glucose,high-density lipoprotein (HDL) cholesterol,low-density lipoprotein (LDL) cholesterol,phosphate,potassium,protein,sodium,triglycerides,urate and urea.Participants were counted in worst case category if their value changed to(low,normal or high),unless there was no change in their category.Participants whose laboratory value category was unchanged(e.g. High to High),or whose value became normal,were recorded in the 'To Normal or No Change' category.Participants were counted twice if the participant had values that changed 'To Low' and 'To High',so the percentages may not add to 100%.Baseline value=latest pre-dose assessment(prior to oral dose) in each treatment period,with a non-missing value,including those from unscheduled visits
Time Frame: Baseline (Day 1: pre-dose) and Up to 50 Days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Participants
  ALT, To Low | 0 | 0
  ALT, To Normal or No Change | 5 | 5
  ALT, To High | 0 | 0
  Albumin, To Low | 0 | 0
  Albumin, To Normal or No Change | 5 | 5
  Albumin, To High | 0 | 0
  ALP, To Low | 0 | 0
  ALP, To Normal or No Change | 5 | 5
  ALP, To High | 0 | 0
  AST, To Low | 0 | 0
  AST, To Normal or No Change | 5 | 5
  AST, To High | 0 | 0
  Bilirubin, To Low | 0 | 0
  Bilirubin, To Normal or No Change | 5 | 5
  Bilirubin, To High | 0 | 0
  Calcium, To Low | 0 | 0
  Calcium, To Normal or No Change | 5 | 5
  Calcium, To High | 0 | 0
  Chloride, To Low | 0 | 0
  Chloride, To Normal or No Change | 4 | 5
  Chloride, To High | 1 | 0
  Cholesterol, To Low | 0 | 0
  Cholesterol, To Normal or No Change | 5 | 5
  Cholesterol, To High | 0 | 0
  Creatinine, To Low | 0 | 0
  Creatinine, To Normal or No Change | 3 | 5
  Creatinine, To High | 2 | 0
  Direct Bilirubin, To Low | 0 | 0
  Direct Bilirubin, To Normal or No Change | 5 | 5
  Direct Bilirubin, To High | 0 | 0
  Globulin, To Low | 0 | 0
  Globulin, To Normal or No Change | 5 | 4
  Globulin, To High | 0 | 1
  Glucose, To Low | 0 | 0
  Glucose, To Normal or No Change | 5 | 5
  Glucose, To High | 0 | 0
  HDL Cholesterol, To Low | 0 | 0
  HDL Cholesterol, To Normal or No Change | 5 | 5
  HDL Cholesterol, To High | 0 | 0
  LDL Cholesterol, To Low | 0 | 0
  LDL Cholesterol, To Normal or No Change | 4 | 5
  LDL Cholesterol, To High | 1 | 0
  Phosphate, To Low | 0 | 0
  Phosphate, To Normal or No Change | 5 | 5
  Phosphate, To High | 0 | 0
  Potassium, To Low | 0 | 0
  Potassium, To Normal or No Change | 5 | 5
  Potassium, To High | 0 | 0
  Protein, To Low | 0 | 0
  Protein, To Normal or No Change | 4 | 5
  Protein, To High | 1 | 0
  Sodium, To Low | 0 | 0
  Sodium, To Normal or No Change | 5 | 5
  Sodium, To High | 0 | 0
  Triglycerides, To Low | 0 | 0
  Triglycerides, To Normal or No Change | 5 | 5
  Triglycerides, To High | 0 | 0
  Urate, To Low | 0 | 0
  Urate, To Normal or No Change | 5 | 5
  Urate, To High | 0 | 0
  Urea, To Low | 0 | 0
  Urea, To Normal or No Change | 5 | 5
  Urea, To High | 0 | 0

55. Secondary Outcome: Number of Participants With Clinically Significant Urinalysis Findings
Description: Urine samples were collected to detect the presence of bilirubin, glucose, ketones, leukocyte esterase, nitrite, occult blood, protein and urobilinogen. Urinalysis also included measurement of specific gravity and potential of Hydrogen (pH). Number of participants with clinically significant urinalysis findings are presented.
Time Frame: Up to 50 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

56. Secondary Outcome: Number of Participants With Worst Case Post Baseline Abnormal 12-Lead Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were recorded with the participants in semi-supine position after 5 minutes rest using an automated ECG machine that measured PR, QRS, QT and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. Data for number of participants with abnormal, not clinically significant (NCS) and Clinically significant (CS) ECG findings for worst case post-Baseline are presented. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Baseline value is defined as the latest pre-dose assessment (prior to the oral dose) in each treatment period, with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1: pre-dose) and Up to 50 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Participants
  Abnormal, NCS | 2 | 3
  Abnormal, CS | 0 | 0

57. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in semi-supine position after 5 minutes rest with a completely automated device. Baseline value is defined as the latest pre-dose assessment (prior to the oral dose) in each treatment period, with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: pre-dose), Day 1 (4 hours) and Day 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Millimeters of mercury (mmHg)
  SBP: Day 1 (4 hours); n= 5, 4: number analyzed (Participants) | 5 | 4
  SBP: Day 1 (4 hours); n= 5, 4 | 3.4 (6.95) | -0.3 (5.38)
  DBP: Day 1 (4 hours); n = 5, 4: number analyzed (Participants) | 5 | 4
  DBP: Day 1 (4 hours); n = 5, 4 | 2.6 (6.19) | 3.0 (3.37)
  SBP: Day 8; n= 5, 5 | 2.8 (5.07) | 3.0 (6.82)
  DBP: Day 8; n= 5, 5 | 2.8 (6.30) | -5.8 (6.98)

58. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in semi-supine position after 5 minutes rest with a completely automated device. Baseline value is defined as the latest pre-dose assessment (prior to the oral dose) in each treatment period, with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: pre-dose), Day 1 (4 hours) and Day 8
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Beats per minute
  Pulse rate: Day 1 (4 hours); n= 5, 4: number analyzed (Participants) | 5 | 4
  Pulse rate: Day 1 (4 hours); n= 5, 4 | -3.8 (7.53) | -2.3 (2.22)
  Pulse rate: Day 8; n= 5, 5 | 8.2 (7.19) | 0.0 (5.29)

59. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in semi-supine position after 5 minutes rest. Baseline value is defined as the latest pre-dose assessment (prior to the oral dose) in each treatment period, with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: pre-dose), Day 1 (4 hours) and Day 8
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Breaths per minute
  Respiratory rate: Day 1 (4 hours); n= 5, 4: number analyzed (Participants) | 5 | 4
  Respiratory rate: Day 1 (4 hours); n= 5, 4 | 0.0 (2.83) | -1.0 (1.15)
  Respiratory rate: Day 8; n= 5, 5 | 0.8 (1.79) | 0.8 (1.10)

60. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature was measured in semi-supine position after 5 minutes rest. Baseline value is defined as the latest pre-dose assessment (prior to the oral dose) in each treatment period, with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: pre-dose), Day 1 (4 hours), 36, 72, 96, 120, 144, 168 hours and Day 8
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Degree Celsius
  Temperature: 4 hours; n= 5, 4: number analyzed (Participants) | 5 | 4
  Temperature: 4 hours; n= 5, 4 | 0.28 (0.259) | 0.38 (0.403)
  Temperature: 36 hours; n= 5, 5 | 0.04 (0.404) | 0.28 (0.383)
  Temperature: 72 hours; n= 5, 5 | 0.24 (0.336) | 0.32 (0.415)
  Temperature: 96 hours; n= 5, 5 | 0.32 (0.421) | 0.08 (0.363)
  Temperature: 120 hours; n= 5, 5 | 0.26 (0.321) | -0.14 (0.329)
  Temperature: 144 hours; n= 5, 5 | 0.08 (0.356) | 0.00 (0.430)
  Temperature: 168 hours; n= 5, 5 | 0.12 (0.277) | 0.08 (0.492)
  Temperature: Day 8; n= 5, 5 | 0.36 (0.385) | 0.16 (0.270)

61. Secondary Outcome: Change From Baseline in Weight
Description: Weight was measured and recorded. Baseline value is defined as the latest pre-dose assessment (prior to the oral dose) in each treatment period, with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: pre-dose) and up to Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | GSK3640254 Tablet + [14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5 | 5
Kilograms | -0.64 (0.792) | -1.10 (0.892)

62. Secondary Outcome: Total Radioactivity in Blood to Plasma Following Administration of Oral Dose of [14C]-GSK3640254
Description: Blood samples were collected at the indicated time points for analysis of total radioactivity in blood to plasma. It was calculated as Radioactivity Concentration in blood (Cb) divided by Radioactivity Concentration in plasma (Cp).
Time Frame: Day 1: 2, 4, 6, 8 and 10 hours
Population: PK Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | [14C]-GSK3640254 Oral Suspension
Number analyzed (Participants) | 5
Ratio
  2 hours | 0.555 (0.0340)
  4 hours | 0.480 (0.0844)
  6 hours | 0.522 (0.0429)
  8 hours | 0.503 (0.0249)
  10 hours | 0.595 (0.164)

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-serious AEs were collected from the start of study treatment up to Day 50.
Description: SAEs and Non-SAEs were reported for the Safety Population which comprised of all participants who received at least one dose of study treatment.
Groups:
- GSK3640254 Tablet+[14C]-GSK3640254 IV: Participants were administered a single oral dose of GSK3640254 200 milligram (mg) (2×100 mg) tablets with a moderate fat meal, followed by an intravenous (IV) infusion of [14C]-GSK3640254 100 micrograms for 1 hour on Day 1 in Treatment Period 1. The treatment periods were separated by a washout period of at least 13 days between oral doses.
- [14C]-GSK3640254 Oral Suspension: Participants were administered a single oral dose of 85 mg [14C]-GSK3640254 as an oral suspension with a moderate fat meal in Treatment Period 2 on Day 1. The treatment periods were separated by a washout period of at least 13 days between oral doses.
Arm/Group | GSK3640254 Tablet+[14C]-GSK3640254 IV | [14C]-GSK3640254 Oral Suspension
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3640254 Tablet+[14C]-GSK3640254 IV (N=5) | [14C]-GSK3640254 Oral Suspension (N=5)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT04507321/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04507321/SAP_001.pdf